CLINICAL TRIAL: NCT05758454
Title: Innovation Project Innovation Project for the Public Sector: Caries-Obesity Prevention in Children by Modifying Risk Behaviors Among Parents With Immigrant Background-COP Study
Brief Title: Caries-Obesity Prevention in Children by Modifying Risk Behaviors Among Parents With Immigrant Background-COP Study
Acronym: COP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oral Health Centre of Expertise in Western Norway (Other)
Collaborators: University of Bergen (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Manal Ibrahim Mustafa Sharafeldin, Researcher, Oral Health Centre of Expertise in Western Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OralHCentre
Record Dates: First submitted 2022-12-09; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Oral Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral health information (Other): Intervention in form of a health/dental health information translated into different native language will be provided for the intervention group
  Interventions: Behavioral: Caries and Obesity Prevention

INTERVENTIONS:
Behavioral: Caries and Obesity Prevention — A culturally adapted oral health education intervention to prevent development of ECC and to improve parental oral health related knowledge and attitudes.
  Other Names: COP

SUMMARY:
Immigrants constitute 18.2 % of the whole population in Norway. Health inequalities were previously reported, and immigrant status has been associated with a high risk of caries and obesity in children. Lack of parental knowledge, poor communication, ethnic and cultural differences are suggested to be reasons for the observed discrepancies. Therefore, research-based knowledge about the social, psycho-social and cognitive factors, that direct health / dental health-related behavior in families with an immigrant background is needed.

Aims The main goal of this project is to assess attitudes and behaviors related to health/oral health among immigrant parents with newborn children (0-6 months). Develop an intervention programs with the aim of increasing the parent's knowledge of the children's oral hygiene/food habits and to evaluate in a follow-up study the effect of intervention on parents' knowledge and attitude with regard to dental caries and obesity.

Methods Parents with immigrant status will be recruited from primary health centers located in the western part of Norway when meeting for children's vaccination. Primary health care centers will be conveniently divided into an intervention and control group. Intervention in form of a health/dental health information translated into different native language will be provided for the intervention group. The control group will receive regular primary care health information. Efficacy of the intervention will be assessed as differences in change scores between intervention and control group regarding parental attitudes, knowledge and behaviors and children's quality of life related to health and oral health, children's body mass index and early childhood caries. Objective of this work are consistent with community needs to eliminate health/social inequalities and it is anticipated that a culturally adapted interventions can be implemented among immigrant families at a moderate cost.

DETAILED DESCRIPTION:
Detailed Description:

Project Plan

Innovation Project Innovation Project for the Public Sector. Innovative intervention: Caries-Obesity Prevention in children by modifying risk behaviors among parents with immigrant background-COP study

Project partner Oral Health Center of Expertise/Western Norway, Hordaland Manal I. Mustafa Sharafeldin Faculty of Medicine and Dentistry University of Bergen Årstadveien 19, Bergen, Norway Anne Nordrehaug Åstrøm Bergen Municipality TkMidtNorge

Rationale of the Study:

In general, evidence of the efficacy of culturally adapted health interventions (interventions that take culture specific factors into account) is scarce. It is assumed that immigrant parents of small children in Bergen may benefit from an early oral health information program that is adapted to their culture, life situation and specific needs as immigrants. An intervention in form of culturally adapted information on oral health to immigrant parents may improve their oral health related knowledge, attitudes and feeding behavior.

As an extension of the intervention study focusing immigrant parents during children's first 18-24 months of life, it is of interest to follow-up this cohort of immigrant parents (i.e., parents from the intervention and control group) and their children from 3 to 5 yrs. of age. Children's primary dentition is fully erupted at the age of 3 yrs. and at that developmental stage children start to attend the public dental health care services for their regular annual check-ups and necessary oral disease treatments. In a follow up of the cohort of immigrant parents and their children it will be possible to assess stability and changes in parental oral health related knowledge and attitudes. Further, it will be beneficial to observe the establishment of children's eating behaviors and long-term impacts on children's dental caries-BMI- and oral health related quality of life status.

AIMS OF THE STUDY General objectives The purpose of this study is to assess oral health related knowledge, attitudes and behavior among immigrant mothers of newborn infants (0-6 months). Further to investigate the potential of a culturally adapted oral health education intervention to prevent development of Early childhood caries (ECC) and to improve parental oral health related knowledge and attitudes. In a prospective follow-up of the cohort of immigrant parents/children (from the intervention study) and a similarly aged control group of Norwegian borne parents /children, we will investigate the changes in parental beliefs related to diet and hygiene from when their children were 3 yrs. until 5 yrs. of age. The development of parental health/oral health related knowledge, children's eating behaviors and the influence on children's subsequent dental caries -, BMI- and oral health related quality of life situation will be compared between immigrants and Norwegian born parents/children.

Objectives

To assess the prevalence and socio-demographic distribution of oral health related knowledge, attitudes and behaviors among parents of infants with immigrant background attending health care centers in Bergen.

To study the efficacy of oral health information program delivered to immigrant mothers of infants aged 0-6 months to improve parental oral health knowledge and to reduce known risk factors for children's caries development at age of 2-3 yrs. old.

In a prospective follow-up study of parents and children with and without immigrant background, compare the development of parental oral health related knowledge and attitudes, children's eating behaviors and the impact on children's caries -, BMI- and oral health related quality of life status at age 5 yrs.

Material & Methods

Study design: This is a cluster randomized controlled intervention followed by a prospective cohort of immigrant parents/ children from the intervention study and a Norwegian born control group.

Immigrant parents for the intervention study will be recruited from health centers located in Bergen. Health centers with high number of parents having immigrant background visiting these centers will be selected. The health centers will be divided into an intervention group receiving a culturally adapted intervention and a control group receiving no culturally adapted intervention. Inclusion criteria: immigrant (born outside Norway) group-parents of non-western origin and having newborn infants (0-6 months) will be included in this study. Non-western background means origin from Eastern Europe, Asia, Africa, South and Central America. Parents of twins will be involved in the study, but only one child conveniently selected will be included. Parents should be able to understand and sign a consent form. Exclusion criteria: newborns with serious congenital defects that expected to adversely affect their oral health will be excluded. The child will be excluded if he/she has situation that required frequent oral health control. The participant will be excluded if they cannot understand and sign a consent form and are not willing to follow the study procedures. All attendees to the respective health centers during the study period will be invited to participate in the study.

The first part of the structured questionnaire- based interview schedules will assess demographics, and socioeconomic status. Demographic data including age, gender, and indicators for socio-economic status: father-mothers' education, occupation. The second part of the questionnaire-based interview will include knowledge about prevention of dental caries and obesity. Attitudes (regular dental visits, tooth cleaning, milk teeth, feeding practice) and Practice (regular dental visits, tooth cleaning, milk teeth, and sugary food intake) assessed among immigrant parents in the baseline (0-6 months after birth) and follow up (18-24 months after birth) of the intervention study as well as in the prospective cohort of immigrants and controls when children are 3 (in 2023) and 5 (in 2025) yrs. of age. An extension of this parental questionnaire, including questions on children's eating behavior and oral health related quality of life will be implemented at 3 and 5 yrs. follow up in the prospective cohort study. The quality of life of children / families with and without immigrant background will be measured using the instrument 'Early Childhood Oral Health Impact Scale (ECOHIS)' including a child and a family part.

The intervention will be provided by project co-workers at an individual level. Eight health centers will be included in the intervention group and 8 health centers will be included as control group without intervention. Intervention will be carried out at baseline 0-6 months after birth. The second round of the intervention will be implemented 6 month later (6-8 month after birth). This will be followed by clinical registration of children's ECC incidence at 18-24 months follow up.

The intervention (oral health information) will be provided in a form of individual presentation in duration of about 30 minutes. Thereafter a practical demonstration of tooth brushing will be provided. Each participant will receive carry home messages in a form of pamphlet containing similar information as in the presentation. The information besides brushing includes information about primary dentition, dietary habits and its effect on prevention of caries and obesity. Further information about bottle feeding and its effect on early childhood caries will be emphasized. Moreover, the importance of regular dental visits will be highlighted. The questionnaire used at baseline will be used again at the end of the study (18-24 month after starting of the study) to evaluate changes in oral health related knowledge- and attitudes.

Prospective cohort study of immigrant parents/children and Norwegian parents/children A prospective follow up study will be carried out between children's age is 3- and 5 years. Immigrant parents/children (from the intervention study) and controls (Norwegian born parents with similarly aged children) will be recruited from the public dental health clinics when they are visiting for routine check-ups of their children at age 3. Immigrant parents /children and controls will be recruited from the same public dental health care clinics. Inclusion criteria: Immigrant parents and their 3 yrs. old children having participated in the interventions study (see inclusion criteria for the intervention study). The control group of Norwegian parents/children are recruited for the first time when children's age is 3 yrs. Exclusion criteria of immigrant parents/children and controls (similar exclusion criteria as stated above in the intervention study).

Also, for the Norwegian control group children with serious congenital defects that expected to adversely affect their oral health will be excluded. The child will be excluded if he/she has situation that required frequent oral health control.

Measurement of parental knowledge and attitudes, children's eating behavior and oral health related quality of life at age 3 and 5 yrs. old: An extension of the parental questionnaire from the intervention study of immigrant parents including questions on children's eating behavior and oral health related quality of life will be implemented at children's aged 3 (in 2023) and 5 yrs. (in 2025) among parents with and without immigrant status. The quality of life of children /families will be measured using the instrument 'Early Childhood Oral Health Impact Scale (ECOHIS)' including a child and a family part. This interview schedule assessing parental knowledge and attitudes and in addition children's eating behaviors will be implemented repeatedly in the prospective follow-up study of immigrant parents /children and control parents/children at children's aged 3 and 5 yrs. Standardized face to face questionnaire-based interviews will be administered at each wave in Norwegian (translator will be considered for those who cannot communicate in Norwegian) by trained interviewers.

Measurement of children's dental caries and BMI status at age 5:

Dental caries in children with and without immigrant background will be assessed by extracting data from dental journals and in terms of dmft (decayed, missed and filled teeth) at 5 yrs. of age. Basic anthropometric measures BMI will be determined according to standardized routines: height (recorded to the nearest centimetre) and body weight (to the nearest 0.5 kg) on lightly dressed children without shoes, and the BMI will be calculated depending on age and sex.

Statistical analysis:

Sample size will be calculated to 200 for each group by using sample size formula for one sided student sample t test. The Statistical package of social sciences (SPSS) version 21 will be used to analyze the data. P value will be set to be 0.05 as a level of significance. Chi-square and dependent sample T tests will be used to assess the difference in categorical and normally distributed continuous variables and to identify possible confounding variables.

The prospective cohort study starting in 2023 will recruit about 200 immigrants parents and their 3 yrs. old children from the intervention study and 200-300 controls for comparison, constituting Norwegian born parents and their 3 yrs. old children. Both groups will be followed prospectively until their children completed 5 yrs. in 2025. Changes in parental knowledge and attitudes and changes in children's eating behavior between 2023 and 2025 as well as the influence on children's caries and BMI status in 2025 will be analyzed using standardized logistic regression analyses. Mixed models to account for the cluster effect in the repeated data.

Ethical and Legal Considerations Ethical approval was obtained (2015/2037/REK vest) from the Regional Ethical Committee (REK), for the intervention part where the efficacy of additional oral health information program delivered to immigrant parents and its impact on subsequent ECC will be investigated the (first part of the Project). The prospective follow up study between children aged 3 to 5 yrs. of age, focusing immigrant parent/children from the intervention study and a new recruited Norwegian born parent/children control groupwhere the parental beliefs will be tracked during the period between 2023 to 2025. In this prospective follow-up study of parents and children with and without immigrant background, the development of parental oral health related knowledge and attitudes, children's eating behaviors and the impact on children's caries -, BMI- and oral health related quality of life situation at age 5 yrs. will be investigated. In the prospective follow up, immigrant parents from the intervention study and the Norwegian controls will sign an informed consent on behalf of themselves and their 3-year-old children.

After completion of the intervention study, this project will be extended with a prospective follow-up study planned to be implemented between 2023 and 2025, including the participants from the intervention study (IM) and a control group of Norwegian parents / children (N) recruited in 2023. Such a follow-up study will make it possible to measure changes in immigrant parents and Norwegian parents' knowledge, attitudes and behaviors across time, establishment of children's eating behavior at age 3 and 5 yrs. Further it will detect the possible influence of parental factors and children's eating behavior on children's caries-, BMI-, and oral health related quality of life situation at 5 yrs. of age. This part is also approve (2015/2037/REK vest) Publication and presentation of the study results The results of this project should be of interest to the scientific community as well as to the professionals, so it is planned to communicate results to these groups through seminars, presentations, meetings and through international publications.

ELIGIBILITY:
Inclusion Criteria:

* Parents having newborn infants (0-6 months) with Non-Western immigrant background

Exclusion Criteria:

* The parents will be excluded if they cannot understand and sign a consent form and are not willing to follow the the clinical trial procedures.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in poor parental knowledge regarding children oral health | Response of parents to the first questionnaire when child is 6 months, and when the child is 24 months.
  The questionnaire applied to the parents before and after cultured adapted informational to compare intervention will be used to measure the change of the parental knowledge. The comparison will be carried out between and within the control and intervention groups.
Change in poor parental behavior regarding children oral health | Response of parents to the first questionnaire when child is 6 months, and when the child is 24 months.
  The questionnaire applied to the parents before and after cultured adapted informational intervention will be used to measure the change of the parental behavior. The comparison will be carried out between and within the control and intervention groups.

SECONDARY OUTCOMES:
Caries increment (Child age 24 months) | Clinical examination when child is 24 months (Duration of clinical examination 15 minutes for each child)
  Clinical examination to measure caries lesions on the upper anterior teeth when the child is 24 months of age. Examination at 6 months is not possible because child at this age has no teeth. The comparison will be carried out between and within the control and intervention groups.
Caries increment (Child age 3 and 5 years old) | Registration of record at child aged 3 and 5 years old (Registration 15-20 minutes for each child)
  Reporting caries increment from child records at the public dental health clinic at age of 3 and 5 years old. The comparison will be carried out between the control (Norwegian parents) and the test (immigrant parents) groups.
Body Mass Index (BMI) (Child age 5 years old) | Response of parents to the first questionnaire when child is 3 years, and when the child is 3 years of age.
  The body mass index of the child will be determined at 5 years of age by measuring the height and the weight of the child. The comparison will be carried out between the control (Norwegian parents) and the test (immigrant parents) groups.
Quality of life of children /families | Response of parents to the first questionnaire when child is 3 years, and when the child is 3 years of age.
  The quality of life of children /families will be measured using the instrument 'Early Childhood Oral Health Impact Scale (ECOHIS)' including a child and a family part. The comparison will be carried out between the control (Norwegian parents) and the test (immigrant parents) groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Berggreen, PhD, Study Director — Oral Health Centre of Expertise in Western Norway
Locations (2):
- Norway (2):
  - Health Centers, Bergen
  - Manal Mustafa, Bergen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reda M, Gwanzura Ottemoller F, Mustafa M. Immigrant parents' perspectives on children's oral health and barriers to a culturally adapted intervention in Norway. Front Oral Health. 2026 Jan 6;6:1726535. doi: 10.3389/froh.2025.1726535. eCollection 2025. PMID 41568138
- [Derived] Reda M, Sen A, Astrom AN, Mustafa M. Effects of an intervention on immigrant parents' knowledge and attitudes toward their children's oral health: A cluster randomized trial in Norway. Eur J Oral Sci. 2025 Feb;133(1):e13037. doi: 10.1111/eos.13037. Epub 2025 Jan 17. PMID 39821537
- [Derived] Reda M, Sen A, Mustafa M. Prevention of caries and obesity in children with immigrant background in Norway- a study protocol for a cluster randomized controlled trial. BMC Oral Health. 2023 Sep 1;23(1):620. doi: 10.1186/s12903-023-03329-9. PMID 37658341